CLINICAL TRIAL: NCT03257202
Title: Cutibacterium Acnes Persists Despite Topical Clindamycin and Benzoyl Peroxide
Brief Title: Topical Treatment and Prevalence of P. Acnes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, George F. Hatch, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS-17-00319
Record Dates: First submitted 2017-08-01; First posted 2017-08-22 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Surgical Site Infection
Keywords: Propionibacterium Acnes; Surgical Site Infection; Shoulder
MeSH Terms: conditions — Surgical Wound Infection | interventions — Clindamycin; Gels; Benzoyl Peroxide; clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control (No Intervention): No topical treatment
- Clindamycin alone (Experimental): topical clindamycin alone using Clindamycin 1% Gel
  Interventions: Drug: Clindamycin 1% Gel
- Benzoyl peroxide alone (Experimental): topical benzoyl peroxide alone using Benzoyl Peroxide 5% Gel
  Interventions: Drug: Benzoyl peroxide 5% gel
- Clindamycin and benzoyl peroxide (Experimental): Topical clindamycin and topical benzoyl peroxide together using BenzaClin 5%-1% Topical Gel
  Interventions: Drug: BenzaClin 5%-1% Topical Gel

INTERVENTIONS:
Drug: Clindamycin 1% Gel — topical clindamycin
  Arms: Clindamycin alone
Drug: Benzoyl peroxide 5% gel — topical benzoyl peroxide
  Arms: Benzoyl peroxide alone
Drug: BenzaClin 5%-1% Topical Gel — Topical clindamycin and benzoyl peroxide together
  Arms: Clindamycin and benzoyl peroxide

SUMMARY:
This study is about preventing surgical site infections of the shoulder. We hope to learn if clindamycin alone, benzoyl peroxide alone, or clindamycin and benzoyl peroxide together can affect growth of Propionibacterium acnes in the dermal layer.

DETAILED DESCRIPTION:
P. acnes are skin pathogens known to cause surgical site infections despite proper preoperative surgical preparation. Lee et al. showed 70% growth rate of P. acnes despite the application of Choraprep prior to sampling. However, this study was limited as it failed to utilize a control group and only investigated one preparatory technique. Meanwhile, there remains to date no study investigating the effect of topical treatments. The purpose of this study is to investigate how specific topical treatments affect growth in the dermal layer. 12 volunteers who are normal volunteers, students, or employees of USC will each receive 4 punch biopsies from their back above the scapular spine, with each biopsy taken from a region of the skin treated with a different topical (topical clindamycin alone, topical benzoyl peroxide alone, topical clindamycin and benzoyl peroxide together, and a control). A 3df overall test of the treatment indicators will test for any differences in positivity for P Acnes among the treatments; pairwise comparisons among the treatments will adjust for multiple comparisons. A two-tailed statistical test will be performed, testing at an alpha of 0.05, and analyses will also be performed based on hemolytic subtypes.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* age > 18

Exclusion Criteria:

* history of antibiotic use in the last month
* active acne on the back
* non-English speakers (the study personnel do not have adequate training to converse and consent in other languages)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George R Hatch, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes Data will be shared as required with the USC Health Sciences Institutional Review Board. Participant data will be coded with coding identifiers kept separately by research personnel only and destroyed upon completion of the study.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Dumville JC, McFarlane E, Edwards P, Lipp A, Holmes A. Preoperative skin antiseptics for preventing surgical wound infections after clean surgery. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003949. doi: 10.1002/14651858.CD003949.pub3. PMID 23543526
- [Background] Mook WR, Garrigues GE. Diagnosis and Management of Periprosthetic Shoulder Infections. J Bone Joint Surg Am. 2014 Jun 4;96(11):956-965. doi: 10.2106/JBJS.M.00402. Epub 2014 Jun 4. PMID 24897745
- [Background] Matsen FA 3rd, Butler-Wu S, Carofino BC, Jette JL, Bertelsen A, Bumgarner R. Origin of propionibacterium in surgical wounds and evidence-based approach for culturing propionibacterium from surgical sites. J Bone Joint Surg Am. 2013 Dec 4;95(23):e1811-7. doi: 10.2106/JBJS.L.01733. PMID 24306704
- [Background] Lee MJ, Pottinger PS, Butler-Wu S, Bumgarner RE, Russ SM, Matsen FA 3rd. Propionibacterium persists in the skin despite standard surgical preparation. J Bone Joint Surg Am. 2014 Sep 3;96(17):1447-50. doi: 10.2106/JBJS.M.01474. PMID 25187583
- [Background] Saltzman MD, Nuber GW, Gryzlo SM, Marecek GS, Koh JL. Efficacy of surgical preparation solutions in shoulder surgery. J Bone Joint Surg Am. 2009 Aug;91(8):1949-53. doi: 10.2106/JBJS.H.00768. PMID 19651954
- [Background] Wright TE, Boyle KK, Duquin TR, Crane JK. Propionibacterium acnes Susceptibility and Correlation with Hemolytic Phenotype. Infect Dis (Auckl). 2016 Oct 9;9:39-44. doi: 10.4137/IDRT.S40539. eCollection 2016. PMID 27773990
- [Background] Hibbard JS. Analyses comparing the antimicrobial activity and safety of current antiseptic agents: a review. J Infus Nurs. 2005 May-Jun;28(3):194-207. doi: 10.1097/00129804-200505000-00008. PMID 15912075
- [Background] Butler-Wu SM, Burns EM, Pottinger PS, Magaret AS, Rakeman JL, Matsen FA 3rd, Cookson BT. Optimization of periprosthetic culture for diagnosis of Propionibacterium acnes prosthetic joint infection. J Clin Microbiol. 2011 Jul;49(7):2490-5. doi: 10.1128/JCM.00450-11. Epub 2011 May 4. PMID 21543562
- Available data/document: Study Protocol: HS-17-00319 — http://istar.usc.edu
- Available data/document: Informed Consent Form: HS-17-00319 — http://istar.usc.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 12 patients received each of the 4 study arms.
Groups:
- All Study Participants: All study participants received all 4 treatments: control, Clindamycin alone, Benzyl peroxide alone, Clindamycin and Benzoyl Peroxide
Period: Overall Study
Arm/Group | All Study Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 1. Negative Control
  2. Topical benzoyl peroxide alone using Benzoyl Peroxide 5% Gel
  3. Topical clindamycin alone using Clindamycin 1% Gel
  4. BenzaClin 5%-1% Topical Gel: Topical clindamycin and benzoyl peroxide together
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 29.4 [26 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Positive Bacterial Growth Culture Per Treatment Arms
Description: Detected presence of growth of Propionibacterium acnes on bacterial culture (bacteria per mL) by treatment arms.
Time Frame: 21 days
Measure: Number; unit: participants
Groups:
- Negative Control: The participants did not receive treatment in this quadrant.
- Benzoyl Peroxide 5% Topical Gel: This quadrant on the participants' backs were treated with Benzoyl Peroxide 5% topical gel
- Clindamycin 1% Topical Gel: This quadrant of the participants' back received Clindamycin 1% topical gel
- Clindamycin 1% Plus Benzoyl Peroxide 5% Topical Gel: This quadrant on the study participants' backs were treated with Clindamycin 1% plus Benzoyl Peroxide 5% topical gel
Arm/Group | Negative Control | Benzoyl Peroxide 5% Topical Gel | Clindamycin 1% Topical Gel | Clindamycin 1% Plus Benzoyl Peroxide 5% Topical Gel
Number analyzed (Participants) | 12 | 12 | 12 | 12
participants | 10 | 12 | 10 | 10

ADVERSE EVENTS:
Time Frame: 24 days
Arm/Group | Control | Clindamycin Alone | Benzoyl Peroxide Alone | Clindamycin and Benzoyl Peroxide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03257202/Prot_SAP_000.pdf